CLINICAL TRIAL: NCT04197167
Title: Mid-Infrared Spectroscopy as a Real Time Diagnostic Tool for Chronic Endometritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0122-19-HYMC
Record Dates: First submitted 2019-12-04; First posted 2019-12-12 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Endometritis; IVF
MeSH Terms: conditions — Endometritis | interventions — Hysteroscopy

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women undergoing hysteroscopy (Experimental): Patients scheduled to undergo hysteroscopy for the evaluation of abnormal bleeding or abnormal cervical or uterine findings.
  Interventions: Procedure: Hysteroscopy; Device: Infrared Spectroscopy

INTERVENTIONS:
Procedure: Hysteroscopy — Diagnostic procedure
Device: Infrared Spectroscopy — This device uses spectral absorption of the tissue taken during hysteroscopy to determine immediate diagnosis of Chronic Endometritis

SUMMARY:
The Investigator propose to develop an in-vitro technique for the measurement and analysis of freshly excised biopsies during hysteroscopy procedure in patients with suspected Chronic Endometritis (CE) condition. Furthermore, the investigator propose to develop a discrimination model between the CE and inflammatory CE types using the measured spectroscopic data from freshly excised biopsies.

DETAILED DESCRIPTION:
It is common practice that, following hysteroscopy, the clinician needs to wait for about two weeks before the results of the histology are returned and the clinical treatment is initiated. In this research, the investigator intent to show that the mid infrared ATR (Assisted Reproductive Treatment) spectroscopy method will provide the physician with sufficient information about the CE inflammation status in a considerably shorter period of time to allow immediate initiation of the appropriate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo hysteroscopy for the evaluation of abnormal bleeding or abnormal cervical or uterine findings.
* Patients scheduled for any histological evaluation including endometrial biopsy, dilatation and curettage (D&C), biopsy/excision of uterine polyp or fibroid or any other cervical or uterine lesion.
* Age 18 and over.

Exclusion Criteria:

* Pregnant women, minors and lack of judgment women will not included
* At the request of the examined woman

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of infrared spectroscopy (ATR-FTIR technique) with routine histopathology | 2 Years
  Using ATR-FTIR technique of impression smears obtained from CE tissue during standard hysteroscopy procedure will provide a new diagnostic tool for fast diagnosis of CE inflammation and thus assist in the clinical decision process leading to assisted reproductive treatment (ART).

CONTACTS AND LOCATIONS:
Overall Officials: Einat Shalom-Paz, Prof, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel